CLINICAL TRIAL: NCT02981992
Title: Observational Study on T Regulatory Cells in Hemodialysis Patients
Brief Title: T Regulatory Cells in Hemodialysis Patients: Observational Study
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Carmelo Libetta, Professor, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 20100014090
Record Dates: First submitted 2016-11-26; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Haemodialysis Complication; Immune Dysfunction
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sample used to evaluate T cell subpopulations
Oversight: Data Monitoring Committee: No

SUMMARY:
In this observational study, the investigators evaluated the Treg number and function in a population of patients undergoing hemodialysis (HD).

In particular, the investigators considered the relationship of Treg cell status with the different HD modalities and clinical parameters.

DETAILED DESCRIPTION:
Patients on hemodialysis (HD) present an elevated risk of cardiovascular disease, cancer and infectious events that may lead to the high morbidity and mortality rate characteristic of this population. Many causes can explain this increased risk, including inflammation that, in turn, might be secondary to dialysis-specific factors, such as contaminated water, dialysis modality and dialysis membranes used for treatment.

In addition to chronic inflammatory, in HD patients is also present a significant alteration of the immune system resulting in chronic lymphocytic infiltration, alteration of T-helper balance (Th1/Th2) etc. The immune response is controlled by very complex mechanisms; it is mediated by interaction between antigen-presenting cells (APC), CD4+ T helper (Th) and T cells CD4+ CD25+ regulatory (Treg), a cell subpopulation of T CD4+ expressing the IL-2 receptor (CD25) and forkhead factor (foxp 3). Treg cells contribute to the maintenance of peripheral tolerance by suppressing the immune response to self-normal or tumor antigens. Treg cells control population's expansion of peripheral cells and suppress the proliferation of Th activated cells. Accessory molecules such as CTLA-4 receptors, CD28 and IL-2 cytokines and IL-6, contribute to the activation and proliferation of Treg cells.

The characterization by flow cytometry of Treg suffered for a lack of specific surface markers. These cells are generally identified on the basis of contemporary expression of molecules CD4 and CD25, but the specificity of these markers is limited, given that the CD25 is also expressed on activated lymphocytes. Recently it has been showed that the expression of Foxp3 gene is a phenomenon strictly linked to the development of regulatory activity of Treg, and so, the extent of the expression of this gene by Real Time PCR is currently considered the most specific Treg marker. There is very poor data on Treg cells function in HD. A recent study shows that in patients on chronic HD, the number of Treg is lower if compared to healthy subjects. Moreover, the Treg cells of patients on HD would present a significant impairment of their function, assessed as the ability to inhibit lymphocyte proliferation.

Those results, however, are affected by the lack of data on the characteristics of the studied patients and the type of dialysis treatment applied. In contrast, a recent study by our group showed that patients on hemodialysis with poor biocompatible membranes have a greater number of circulating Treg compared with healthy controls matched for age and sex.

Given the absence of other data, it still remains to investigate the actual significance and function of Treg in HD, considering that Treg status might potentially affect the immune response.

Therefore, the purpose of this study was to evaluate the structure and function of Treg cells in patients undergoing HD, also considering their relationship with the different HD modalities and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spKt/V ≥ 1,2

Exclusion Criteria:

* Cancer
* Pregnant or breastfeeding
* Sepsis
* Kidney or other organ transplant
* Major cardiovascular events in the previous 3 months
* Patients unable to understand or interdicted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total number of 30 prevalent patients undergoing chronic renal replacement terapy with hemodialysis (HD) has been included in the evaluation. The study duration was 12 months, with a check of the number and function of Treg every 3 months.
  During the study patients were subjected to dialysis and farmacology treatment as usual, without any alteration linked specifically to this protocol. The number and function of Treg were measured as a percentage of CD4+CD25bright+pre-dialysis in the last week of each third month of the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Treg number | Assessment of Treg number at basal control and then every 3 months for a total study period of 12 months
  Assessment of the number of Treg by flow cytometry.

SECONDARY OUTCOMES:
Treg function | Assessment of Treg function at basal control and then every 3 months for a total study period of 12 months
  Evaluation of Treg function by measuring the ability to inhibit cell proliferation in the context of a mixed lymphocyte reaction.
Effect of dialysis modality | Analysis of the number and function of Treg cells in function of the type of dialysis treatment at basal control and then every 6 months for a total study period of 12 months
  Evaluation of the number and function of Treg cells before and after dialysis (by flow cytometry and in vitro experiments), as a function of the type of dialysis treatment by use of multivariate regression models

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Libetta, Prof, Principal Investigator — Fondazione Policlinico "San Matteo", Pavia- Italy
Locations (1):
- Fondazione Policlinico "San Matteo", Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hendrikx TK, van Gurp EA, Mol WM, Schoordijk W, Sewgobind VD, Ijzermans JN, Weimar W, Baan CC. End-stage renal failure and regulatory activities of CD4+CD25bright+FoxP3+ T-cells. Nephrol Dial Transplant. 2009 Jun;24(6):1969-78. doi: 10.1093/ndt/gfp005. Epub 2009 Feb 4. PMID 19193737
- [Background] Sewgobind VD, van der Laan LJ, Kho MM, Kraaijeveld R, Korevaar SS, van Dam T, Ijzermans JN, Weimar W, Baan CC. Characterization of rabbit antithymocyte globulins-induced CD25+ regulatory T cells from cells of patients with end-stage renal disease. Transplantation. 2010 Mar 27;89(6):655-66. doi: 10.1097/TP.0b013e3181c9cc7a. PMID 20164820
- [Background] Sharif MR, Chitsazian Z, Moosavian M, Raygan F, Nikoueinejad H, Sharif AR, Einollahi B. Immune disorders in hemodialysis patients. Iran J Kidney Dis. 2015 Mar;9(2):84-96. PMID 25851286
- [Background] Uda S, Mizobuchi M, Akizawa T. Biocompatible characteristics of high-performance membranes. Contrib Nephrol. 2011;173:23-29. doi: 10.1159/000328941. Epub 2011 Aug 8. PMID 21865772
- [Result] Libetta C, Esposito P, Sepe V, Portalupi V, Margiotta E, Canevari M, Dal Canton A. Dialysis treatment and regulatory T cells. Nephrol Dial Transplant. 2010 May;25(5):1723-7. doi: 10.1093/ndt/gfq055. Epub 2010 Feb 15. No abstract available. PMID 20157169
- [Derived] Sepe V, Gregorini M, Rampino T, Esposito P, Coppo R, Galli F, Libetta C. Vitamin e-loaded membrane dialyzers reduce hemodialysis inflammaging. BMC Nephrol. 2019 Nov 15;20(1):412. doi: 10.1186/s12882-019-1585-6. PMID 31729973